CLINICAL TRIAL: NCT01394874
Title: Can Computer-based Telephone Counseling Improve Long-term Adherence to Strength Training in Elders With Knee Osteoarthritis (OA)?
Brief Title: Can Computer-based Telephone Counseling Improve Long-term Adherence to Strength Training in Elders With Knee OA?
Acronym: BOOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H133B100003-2
Record Dates: First submitted 2011-06-21; First posted 2011-07-15 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telephone-linked Communication (TLC) (Experimental): This group will receive the computer-based telephone counseling.
  Interventions: Behavioral: TLC
- Control (No Intervention): This is the control group. They will receive the exercise class, however, they will not receive the telephone counseling.

INTERVENTIONS:
Behavioral: TLC — Computer-based telephone linked communication will be used to counsel subjects to adhere to their exercise program over time.
  Arms: Telephone-linked Communication (TLC)

SUMMARY:
The purpose of this research is to determine whether computer-based telephone counseling will improve adherence to strength training in a population of elders with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee (ICD-9 Code of 715.16, 715.09 or 715.9)
* lives within interstate 95
* age 55 or older
* English speaking

Exclusion Criteria:

* Stroke or heart attack in last 3 months
* Treatment for cancer
* Severe systemic disease
* Medical condition that limits physical activity
* Inflammatory arthritis
* Plans for knee replacement
* Dementia or inability to follow exercise instructions and TLC system

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
Self-report measure of exercise adherence over the last 3-months on a numeric rating scale | 24 month
  Exercise adherence was assessed by the single self-report item "How would you rate your level of adherence to the prescribed BOOST exercise program, over the last 3 MONTHS?" Participants selected a number from 0 (not at all) to 10 (completely as instructed). Higher scores reflect better adherence.

SECONDARY OUTCOMES:
24 -month change in self-report of pain and function using the WOMAC index | post the 1-month exercise class, 24 months
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy domestic duties, light domestic duties Responses to individual questions [between 0 (extreme) and 4 (None)] are summed to a raw score ranging from 0 (worst) to 96 (best) and then normalized to a WOMAC Score of between 0 (worst) to 100 (best). The difference in pain and function subscale values between the measures following the exercise class and the 24-month follow-up were used for secondary outcomes.
Quadriceps strength | Change in quadriceps strength from baseline to 24 months.
  Isokinetic quadriceps strength will be assessed with a Biodex
Timed Physical Function tasks | Change in timed physical function task over 24 months
  Timed physical function tasks will include a timed get up and go, timed stair ascent and descent, and a 5 and 10 chair stand time. We will examine the association of adherence, as a dichotomous and continuous variable, to change in timed physical function using logistic and linear regression, respectively.
Exercise quality | Average measure of exercise quality over 24 months
  The outcome will be assessed at the end of the 24 month follow-up period as the number of calendar periods (1 month per calendar period) that the participant exercises at least half the number of prescribed sessions (a minimum of 6 out of 12 over a 4 week period) with the agreed upon level of intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Baker, PhD, Principal Investigator — Boston University Charles River Campus
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baker K, LaValley MP, Brown C, Felson DT, Ledingham A, Keysor JJ. Efficacy of Computer-Based Telephone Counseling on Long-Term Adherence to Strength Training in Elderly Patients With Knee Osteoarthritis: A Randomized Trial. Arthritis Care Res (Hoboken). 2020 Jul;72(7):982-990. doi: 10.1002/acr.23921. PMID 31074576
- [Derived] Chang FH, Jette AM, Slavin MD, Baker K, Ni P, Keysor JJ. Detecting functional change in response to exercise in knee osteoarthritis: a comparison of two computerized adaptive tests. BMC Musculoskelet Disord. 2018 Jan 23;19(1):29. doi: 10.1186/s12891-018-1942-9. PMID 29361920